CLINICAL TRIAL: NCT06227364
Title: PRE3 PRE-CUBE. PREdiction, PREvention, PREdisposition: Applications in Neurology and Endocrinology
Brief Title: Prediction, Prevention, Predisposition: Applications in Neurology and Endocrinology
Acronym: PRECUBE2022
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Centro Neurolesi Bonino Pulejo (Other)
Responsible Party: Sponsor
Other Study IDs: PRECUBE2022
Record Dates: First submitted 2024-01-09; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-07

CONDITIONS: Dementia; Mild Cognitive Impairment
MeSH Terms: conditions — Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MCI patients: patients with mild cognitive impairment submitted to Magnetic Resonance, neuropsychological evaluation, neurological assessment
  Interventions: Diagnostic Test: MCI patients
- Metabolic patients: patietns with obesity and metabollic dysfunction submitted to haematological tests, psychological and neuropsychological evaluations and endocrinology assessment
  Interventions: Diagnostic Test: metabolic patients

INTERVENTIONS:
Diagnostic Test: MCI patients — patients with mild cognitive impairment submitted to Magnetic Resonance, neuropsychological evaluation, neurological assessment
  Groups: MCI patients
Diagnostic Test: metabolic patients — patients with obesity and metabolic dysfunction submitted to haematological tests, psychological and neuropsychological evaluation and endocrinologu assessment
  Groups: Metabolic patients

SUMMARY:
This project aims to introduce solutions for strengthening the management capabilities of two types of patients, in terms of care and prevention. Specifically, it is aimed at neurological patients with mild or minor neurocognitive decline (Mild Cognitive Impairment, MCI) and endocrinological patients diagnosed with obesity. The study want to enhance the predictive capacity of the care process management system through an Artificial Intelligence (AI) system. All patients diagnosed with MCI and obesity who, within 30 months, will be referred to the Neurology and Endocrinology clinics of the IRCCS Centro Neurolesi Bonino-Pulejo in Messina will be evaluated.

Study design

Patients will not be subjected to any procedure that goes beyond normal clinical practice; the clinical and neuropsychological variables that will be collected for the study are those that are commonly collected in normal clinical practice. All patients diagnosed with MCI and obesity who, within 30 months, will be referred to the Neurology and Endocrinology clinics of the IRCCS Centro Neurolesi Bonino-Pulejo in Messina will be evaluated.

All patients will undergo clinical, neuropsychological and psychological evaluation at the beginning (baseline T0), at the end (T1) and after ... months from the end of treatment (follow up T2).

DETAILED DESCRIPTION:
This project aims to introduce solutions for strengthening the management capabilities of two types of patients, in terms of care and prevention. Specifically, it is aimed at neurological patients with mild or minor neurocognitive decline (Mild Cognitive Impairment, MCI) and endocrinological patients diagnosed with obesity. The study want to enhance the predictive capacity of the care process management system through an Artificial Intelligence (AI) system. All patients diagnosed with MCI and obesity who, within 30 months, will be referred to the Neurology and Endocrinology clinics of the IRCCS Centro Neurolesi Bonino-Pulejo in Messina will be evaluated.

Study design

Patients will not be subjected to any procedure that goes beyond normal clinical practice; the clinical and neuropsychological variables that will be collected for the study are those that are commonly collected in normal clinical practice. All patients diagnosed with MCI and obesity who, within 30 months, will be referred to the Neurology and Endocrinology clinics of the IRCCS Centro Neurolesi Bonino-Pulejo in Messina will be evaluated.

All patients will undergo clinical, neuropsychological and psychological evaluation at the beginning (baseline T0), at the end (T1) and after ... months from the end of treatment (follow up T2).

ELIGIBILITY:
Inclusion Criteria:

For MCI patients:

Patients aged between 18 and 80 years; Clinical and instrumental diagnosis of MCI, according to the normal clinical practice adopted; Written informed consent obtained from the patient;

For Metabolic patients:

Age: >18 years BMI > 30 kg/m²

Willingness to follow requests as per protocol, including:

Signing an informed consent. Participation in scheduled follow-up visits. Carrying out instrumental and laboratory tests

Exclusion Criteria:

For MCI patients:

age under 40 other concomitant neurological and/or psychiatric condition drug abuse unstable clinical conditions requiring acute hospitalization.

For Metabolic patients:

unstable clinical conditions requiring acute hospitalization. associated serious pathologies and/or with reduced life expectancy, including renal failure under dialysis treatment, liver cirrhosis, malignant neoplasms, NYHA class III-IV heart failure, chronic respiratory failure under oxygen therapy.

psychological or psychiatric conditions that may reduce study cooperation.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: N 100 patients diagnosed with MCI and N 100 patients with BMI > 30 kg/m² with or without comorbidities, coming from the external basin, family doctors or other specialists, will be recruited at the Neurology and Endocrinology clinics of the IRCCS Centro Neurolesi Bonino Pulejo of Messina.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2025-01-21 (Estimated)

PRIMARY OUTCOMES:
the creation of predictive algorithms capable of calculating the risk of onset and/or staging of neurodegenerative and metabolic pathologies | 1 hour
  The project has as its primary objective the creation of predictive algorithms capable of calculating the risk of onset and/or staging of neurodegenerative and metabolic pathologies, with the aim of identifying potential targets of subjects at risk of developing such diseases, in the context of patient enrollment, as per normal clinical practice, on an outpatient basis, at our IRCCS.

SECONDARY OUTCOMES:
Evaluate the effectiveness of the therapeutic path and define the outcomes of the treatment plan for these types of patients | 1 hour
  Consider the macro-tasks relating to Taking Charge, Activation of the therapeutic, care and rehabilitation plan as well as the activation of care and follow-up services. With these macro-tasks, through an analysis of the data, it will be possible to carry out an evaluation of the effectiveness of the treatment path envisaged for the patient, identify the treatment process that follows the adopted PDTA (taking charge, evaluation, monitoring and follow-up up) and define the outcomes of the treatment plan for these types of patients, promoting a correct diagnostic classification and an effective therapeutic intervention aimed at managing comorbidities and improving the patients' quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Centro Neurolesi Bonino Pulejo, Messina, Italy